CLINICAL TRIAL: NCT05656209
Title: Lactobacillus Acidophilus Improves the Prognosis (Cognitive Function) of Patients With Ischemic Cerebrovascular Disease After Surgery: a Prospective Randomized Controlled Study
Brief Title: LA Improves the Prognosis of Patients With ICVD After Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huaqiu Zhang (Other)
Responsible Party: Sponsor-Investigator, Huaqiu Zhang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13419632963
Record Dates: First submitted 2022-08-19; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Ischemia; Cerebrovascular; Cognitive Impairment
MeSH Terms: conditions — Cerebral Infarction; Cognitive Dysfunction | interventions — Lacteol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The patient received conventional care after surgery, with no other interventions.
- LA treatment group (Experimental): The patient received conventional treatment and Lactobacillus acidophilus treatment for three months after surgery.
  Interventions: Dietary Supplement: Lactobacillus acidophilus

INTERVENTIONS:
Dietary Supplement: Lactobacillus acidophilus — Lactobacillus acidophilus solid drink (pure bacteria, food grade, JYLA-191, Shandong Zhongke Jia-yi Biological Engineering Co., LTD.), 3G (containing 2*10^10CFU), twice a day, once in the morning and once in the evening, 1 bag each time, by drinking water, direct oral intake, 1 month/course, continuous use for three courses.
  Arms: LA treatment group

SUMMARY:
Ischemic cerebrovascular disease will cause serious harm to the life and safety of patients, and the treatment prognosis is poor. Numerous clinical trials have demonstrated that probiotics can improve cognitive function in people under multimodal. We have previously found that Lactobacillus acidophilus administration could improve cognitive impairment in MCAO and BCAS mice. Therefore, Based on the above research background and the basis of previous studies, we believe that the administration of Lactobacillus acidophilus solid drink (pure Lactobacillus acidophilus strain) can improve the cognitive function of patients with cerebral ischemia through the "brain-gut axis".

DETAILED DESCRIPTION:
Ischemic cerebrovascular disease, as a common form of stroke, is one of the main causes of global morbidity and mortality. The mortality rate of this disease is relatively high, and the treatment prognosis is poor, which will cause serious harm to the life and safety of patients. The optimal treatment for ischemic cerebrovascular disease is still unclear, and the effects of different treatments are still controversial. Therefore, it is of great clinical significance to explore a safe and simple adjuvant treatment method to help patients recover their nervous system function faster and better.

At present, numerous clinical trials have demonstrated that probiotics can improve cognitive function in people under multimodal. Adding intestinal probiotics can improve the intestinal flora distribution, and significantly improve cognitive function in elderly patients with mild cognitive impairment and prevention of brain atrophy. Lactobacillus acidophilus is rich in short chain fatty acids (SCFA). Clinical studies have shown that SCFA levels are negatively correlated with the severity and prognosis of ischemic stroke. Numerous studies have demonstrated that the intestinal supply short chain fatty acids can improve cognitive function, in the middle cerebral artery occlusion (MCAO) induced by acute cerebral ischemia model, rich in the intestines of SCFA can cure acute cerebral ischemia in mice induced by nerve injury. More importantly, in mice with acute cerebral ischemia induced by middle cerebral artery occlusion (MCAO) and chronic cerebral ischemia caused by bilateral common carotid artery stenosis (BCAS), we have previously found that mice have cognitive impairment, accompanied by intestinal flora dysregulation.

Lactobacillus acidophilus administration has a significant effect on improving cognitive function. Based on the above research background and the basis of previous studies, the researchers believe that the administration of Lactobacillus acidophilus solid drink (pure Lactobacillus acidophilus strain) can improve the cognitive function of patients with cerebral ischemia through the "brain-gut axis", and increase the reliability and scope of revascularization, and ultimately improve the prognosis of patients with ischemic cerebrovascular disease.

ELIGIBILITY:
Inclusion Criteria:

1. 35-60 years old;
2. Diagnosed as ischemic cerebrovascular disease, mild to moderate symptoms, can independently complete the neuropsychological test;
3. No previous operation history;
4. The modified Rankin scale score was 0 or 1;
5. Carotid artery ischemic symptoms ≤3 months before treatment;
6. Surgical treatment;

Exclusion Criteria:

1. Previous dementia;
2. hearing or visual impairment;
3. drugs that may or are known to affect cognitive abuse;
4. alcohol addiction;
5. Diagnosis of depression, schizophrenia and other mental diseases;
6. MRI showed severe cerebral infarction;
7. Patients with Lactobacillus acidophilus allergy.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 236 (Estimated)
Dates: Start 2022-12-18 (Estimated); Primary Completion 2022-12-18 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Mini-mental State Examination (MMSE, 0-30) scale | Three months.
  Higher scale scores mean better cognitive function.
Montreal Cognitive Assessment (MoCA, 0-30) scale | Three months.
  Higher scale scores mean better cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Huaqiu Zhang, PhD, Study Director — Tongji Hospital

IPD SHARING:
Plan to Share IPD: No